CLINICAL TRIAL: NCT06186973
Title: Fetal Assessment of the Myocardium and Evaluation of the Neonate
Acronym: FAME-n
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Anne Lee Solevåg, Consultant physician, Oslo University Hospital
Other Study IDs: 28911
Record Dates: First submitted 2023-12-01; First posted 2024-01-02 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Newborn Asphyxia; Hemodynamic Instability; Myocardium; Ischemic; Fetal Distress; Labor Pain
MeSH Terms: conditions — Asphyxia Neonatorum; Coronary Artery Disease; Fetal Distress; Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Umbilical cord blood - preferably arterial Maternal arterial blood gases from the radial artery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No maternal epidural labor analgesia: Term infants monitored with cardiotocography with ST-segment analysis (STAN) during labour: No maternal epidural labor analgesia
  Interventions: Other: Monitoring with Neobeat heart rate meter; Other: Maternal arterial blood gases; Other: Amniotic fluid lactate
- With maternal epidural labor analgesia: Term infants monitored with cardiotocography with ST-segment analysis (STAN) during labour: With maternal epidural labor analgesia
  Interventions: Other: Monitoring with Neobeat heart rate meter; Other: Maternal arterial blood gases; Other: Amniotic fluid lactate

INTERVENTIONS:
Other: Monitoring with Neobeat heart rate meter — At the designated time for cord clamping as per clinical indication, a 10 cm segment of the umbilical cord will be double-clamped and 5 ml of preferably arterial blood will be obtained.
  In infants brought to the resuscitation table, six ECG electrodes will be placed on the skin and cardiac output will be measured with a hemodynamic monitor (PhysioFlow®) for at least 10 min, or until the end of resuscitation/stabilization.
  Other Names: Umbilical cord blood withdrawal and Monitoring with impedance cardiography
Other: Maternal arterial blood gases — Arterial blood gases will be drawn from a radial artery line and analyzed at the end of a contraction at pre-specified time points during labor.
Other: Amniotic fluid lactate — Amniotic fluid will be collected (2mL) and analyzed at pre-specified time points after rupture of the membranes.

SUMMARY:
FAME-n aims to improve perinatal care by introducing new approaches to fetal and neonatal heart assessment. Better identification of high-risk deliveries requiring intervention will reduce perinatal asphyxia-related illness and death. Neonatal hemodynamics may be improved by early detection of instability of the heart and circulation. Innovative use of technology enables characterization of normal and abnormal cardiovascular transition in a significantly larger number of fetuses and newborn infants than what was previously possible. The methods used may have broad generalizability and applicability in perinatal, neonatal and pediatric medicine.

In September 2023, the project was expanded with an obstetric arm called Epidural analgesia: Fetal Oxygenation and Maternal Oxygenation (Epi-FOMO). In Epi-FOMO, the relationship between maternal breathing and arterial blood gases during labour, and umbilical cord blood gases and neonatal outcomes (as specified in FAME-n) will be investigated.

DETAILED DESCRIPTION:
Among the millions of infants with various degrees of perinatal asphyxia each year, the question how to identify those that without supportive measures will die or develop brain injury remains unanswered. The very small population of infants with severe compromise and requiring advanced delivery room resuscitation and therapeutic hypothermia represents only the tip of the iceberg of infants that die or survive with neurological impairment. Thus, the majority of infants with a poor outcome are difficult to distinguish from those with a healthy survival. This challenge persists because currently used markers of perinatal asphyxia are inadequate and unspecific. Better methods to diagnose and monitor hypoxia-ischemia are called for.

The project will characterize in detail both normal and failed (resulting in perinatal asphyxia) transition from fetal to neonatal life. We will study the fetal/neonatal heart throughout perinatal transition, as a continuum and a single physiological entity. This cross-disciplinary approach is groundbreaking as it challenges current clinical practice, knowledge and research. Innovative use of existing technology contributes to further exploring the heart to provide prognostic information and guide supportive therapy.

The target group is fetuses and newborn infants with mild to moderate perinatal asphyxia, i.e., "uncomplicated" infants at birth that later die or develop brain injury.

Our research question is whether immediate neonatal electrocardiogram (ECG) corresponds to fetal ECG as monitored by cardiotocography (CTG) with ST-segment analysis (STAN), and whether neonatal ECG morphology differentiates between infants with mild to moderate perinatal asphyxia and healthy infants. Umbilical cord blood biomarkers, clinical outcomes and secondarily, cardiac output will be used to answer the research question.

For the Epi-FOMO study arm - maternal blood samples during labor will be drawn from an arterial line. The Epi-FOMO participants are a subset of those included in FAME-n, and we will include an equal number of delivering women with and without epidural analgesia. The hypothesis is that epidural analgesia affects maternal breathing and gas exchange, which in turn affects fetal gas exchange and the condition of the newborn infant. We believe that measurement of amniotic fluid lactate during labor may serve as "proof of concept" that maternal respiration during labor modifies the risk of perinatal asphyxia.

ELIGIBILITY:
Inclusion Criteria:

Women admitted for labor and newborn infants will be included after written consent from both parents (if applicable). The final inclusion criterion is that CTG with STAN is used for fetal surveillance at clinician's discretion.

Exclusion Criteria:

Perinatal asphyxia fulfilling the criteria for therapeutic hypothermia, major malformations and stillbirth, known chromosomal anomalies or congenital heart defects other than a patent ductus arteriosus.

Ages: 0 Hours to 1 Hour | Sex: All
Age Groups: Child
Study Population: STAN is used in combination with CTG in fetuses >36 weeks of gestation. Thus, the study population will only include infants born with a gestational age >36 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2030-11-13 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal ECG | From birth until 10 minutes of age
  Blindly categorized neonatal ECG
Cardiac enzymes | At the designated time for cord clamping as per clinical indication
  Umbilical cord blood cardiac enzymes: Creatine kinase (CK)-MB and troponin T
Cardiac output | From birth at least until 10 minutes of age
  Cardiac output
STAN | 10 minutes prior to delivery
  Blindly categorized STAN ECG raw data

SECONDARY OUTCOMES:
Autonomic function | At the designated time for cord clamping as per clinical indication
  Umbilical cord blood metanephrines

OTHER OUTCOMES:
Maternal arterial blood gases | Four times during 1st stage of labor, during pushing and after delivery, maximum duration 24 hours of total labor time
  Oxygen partial pressure (pO2) and carbondioxide partial pressure (pCO2)
Amniotic fluid lactate | Four times during 1st stage of labor, and during pushing, maximum duration 24 hours of total labor time
  Analyzed in 2mL amniotic fluid

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Waldum, PhD, Principal Investigator — Oslo University Hospital; Anne Lee Solevåg, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided